CLINICAL TRIAL: NCT00387764
Title: An Open-label Extension Study to Assess the Safety and Efficacy of Pazopanib in Subjects With Renal Cell Carcinoma Previously Enrolled on Protocol VEG105192
Brief Title: Extension Study to VEG105192 to Assess Pazopanib in Patients With Advanced/Metastatic Renal Cell Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEG107769
Record Dates: First submitted 2006-10-12; First posted 2006-10-13 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2014-01-14 (Estimated); Status verified 2013-10

CONDITIONS: Carcinoma, Renal Cell
Keywords: renal cell carcinoma; pazopanib; anti-angiogenic therapy; open label
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

ARMS (1):
- pazopanib arm (Experimental): This was a single arm study, therefore no control arm.
  Interventions: Drug: pazopanib

INTERVENTIONS:
Drug: pazopanib — 800 mg daily dosing continously until progression

SUMMARY:
This is an open-label, international, multi-center study designed to provide access to pazopanib for subjects who have been enrolled in the Phase III renal cell carcinoma study (VEG105192) and have progressed on placebo. Subjects will receive 800 mg pazopanib once daily. The study treatment will continue until subjects experience disease progression, unacceptable toxicity, withdrawal of consent, or death. The primary objective of the study is to evaluate the safety and tolerability of pazopanib for the treatment of renal cell carcinoma. The secondary objectives of the study are to assess response rate (defined as complete response or partial response), progression-free survival, and overall survival. Response rates will be collected per investigator assessment (no central review). Subjects will have a CT/MRI scan every 6 weeks until week 24 and every 12 weeks thereafter.

ELIGIBILITY:
Inclusion criteria:

* Progressed from VEG105192 study treatment
* Patient's VEG105192 was placebo
* Baseline has good organ function

Exclusion criteria:

* No brain metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-09; Primary Completion 2009-12 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (50):
- Argentina (5):
  - GSK Investigational Site, Capital Federal, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Quilmes
  - GSK Investigational Site, San Miguel de Tucumán
- Australia (3):
  - GSK Investigational Site, Waratah, New South Wales
  - GSK Investigational Site, Hobart, Tasmania
  - GSK Investigational Site, Heidelberg, Victoria
- Austria (2):
  - GSK Investigational Site, Salzburg
  - GSK Investigational Site, Vienna
- Brazil (2):
  - GSK Investigational Site, Belo Horizonte, Minas Gerais
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
- Chile (2):
  - GSK Investigational Site, Viña del Mar, Región de Valparaíso
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- GSK Investigational Site, Beijing, China
- Czechia (3):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Chomutov
  - GSK Investigational Site, Prague
- GSK Investigational Site, Tartu, Estonia
- GSK Investigational Site, Rome, Lazio, Italy
- GSK Investigational Site, Riga, Latvia
- Lithuania (2):
  - GSK Investigational Site, Kaunas
  - GSK Investigational Site, Vilnius
- New Zealand (2):
  - GSK Investigational Site, Christchurch
  - GSK Investigational Site, Wellington
- Pakistan (2):
  - GSK Investigational Site, Karachi
  - GSK Investigational Site, Lahore
- Poland (3):
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Olsztyn
- Russia (8):
  - GSK Investigational Site, Chelyabinsk
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Omsk
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- GSK Investigational Site, Bratislava, Slovakia
- South Korea (2):
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Songpa-gu, Seoul
- Tunisia (3):
  - GSK Investigational Site, Sfax
  - GSK Investigational Site, Sousse
  - GSK Investigational Site, Tunis
- Ukraine (3):
  - GSK Investigational Site, Donetsk
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Kyiv
- United Kingdom (3):
  - GSK Investigational Site, Bebington, Wirral
  - GSK Investigational Site, Belfast, Northern Ireland
  - GSK Investigational Site, Manchester

RESULTS

PARTICIPANT FLOW:
Groups:
- Pazopanib 800 mg: Participants received pazopanib 800 milligrams (mg) once daily.
Period: Overall Study
Arm/Group | Pazopanib 800 mg
Started | 80
Completed | 49 (Participants completed treatment (until disease progression), but may not have completed the study.)
Not Completed | 31
Not completed — Adverse Event | 12
Not completed — Withdrawal by Subject | 8
Not completed — Sponsor Terminated Study | 1
Not completed — Physician Decision | 1
Not completed — Other | 2
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.5 (10.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 61
Race/Ethnicity, Customized [Number; unit: participants]
  Central/South Asian Heritage (HER) | 2
  Japanese/East Asian HER/South East Asian HER | 10
  White | 68

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE) or Serious Adverse Event (SAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in other situations.
Time Frame: From Baseline to Follow-up (up to 6.230 years)
Population: All Treated Participants (ATP) Population: all enrolled participants who received at least one dose of open-label investigational product
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants
  Any AE | 78
  Any SAE | 27

2. Primary Outcome: Number of Participants With Any Adverse Event (Serious and Non-serious) of the Indicated Severity, Per National Cancer Institute (NCI) Common Terminology Criteria in Adverse Events (CTCAE)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is defined as any untoward medical occurrence that, at any dose: results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; or is a congenital anomaly/birth defect. Medical or scientific judgment should be exercised in other situations. Adverse events were graded for severity according to the NCI CTCAE, version 3.0: Grade 1, mild; Grade 2, moderate; Grade 3 (G3), severe; Grade 4 (G4), life-threatening or disabling; Grade 5, death.
Time Frame: From Baseline to Follow-up (up to 6.230 years)
Population: ATP Population
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants
  Grade 1 | 12
  Grade 2 | 33
  Grade 3 | 22
  Grade 4 | 7
  Grade 5 | 4

3. Primary Outcome: Number of Participants With Adverse Events Related to Investigational Product
Description: An adverse event (AE) is defined as any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. The investigator assessed relatedness between the AE and the investigational product.
Time Frame: From Baseline to Follow-up (up to 6.230 years)
Population: ATS Population
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants | 70

4. Primary Outcome: Median Time on Investigational Product
Description: The time on investigational product (including dose interruptions) is defined as the difference between the date of the last dose of investigational product and the date of the first dose of investigational product plus one.
Time Frame: From Baseline to investigational product discontinuation (up to 6.230 years)
Population: ATS Population
Measure: Median (Inter-Quartile Range); unit: Months
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
Months | 9.7 [3.5 to 20.2]

5. Primary Outcome: Number of Participants With the Indicated Worst-case Toxicity Grade Increase From Baseline for the Indicated Clinical Chemistry Parameters at Any Time Post-Baseline
Description: Clinical chemistry parameters were summarized according to NCI CTCAE, version 4.0: Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling; Grade 5, death. Data are presented for only those parameters for which an increase from Baseline occurred. Clinical chemistry parameters included: alkaline phosphatase (ALP), alanine amino transferase (ALT), aspartate amino transferase (AST), total bilirubin (TB), calcium (hypercalcemia and hypocalcemia), creatinine, glucose (hyperglycemia and hypoglycemia), potassium (hyperkalemia and hypokalemia), magnesium (hypermagnesemia and hypomagnesemia), sodium (hypernatremia and hyponatremia), and phosphate.
Time Frame: From Baseline to investigational product discontinuation (up to 6.230 years)
Population: ATS Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed for different parameters, so the overall number of participants analyzed reflects everyone in the ATS Population.
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants
  ALP, any grade increase, n=77 | 26
  ALP, increase to Grade 3, n=77 | 2
  ALP, increase to Grade 4, n=77 | 0
  ALT, any grade increase, n=78 | 39
  ALT, increase to Grade 3, n=78 | 5
  ALT, increase to Grade 4, n=78 | 1
  AST, any grade increase, n=78 | 43
  AST, increase to Grade 3, n=78 | 5
  AST, increase to Grade 4, n=78 | 1
  Creatinine, any grade increase, n=77 | 26
  Creatinine, increase Grade 3, n=77 | 0
  Creatinine, increase Grade 4, n=77 | 0
  Hypercalcemia, any grade increase, n=71 | 14
  Hypercalcemia, increase to Grade 3, n=71 | 1
  Hypercalcemia, increase to Grade 4, n=71 | 1
  Hyperglycemia, any grade increase, n=77 | 46
  Hyperglycemia, increase to Grade 3, n=77 | 1
  Hyperglycemia, increase to Grade 4, n=77 | 0
  Hyperkalemia, any grade increase, n=77 | 28
  Hyperkalemia, increase to Grade 3, n=77 | 4
  Hyperkalemia, increase to Grade 4, n=77 | 1
  Hypermagnesemia, any grade increase, n=77 | 15
  Hypermagnesemia, increase to Grade 3, n=77 | 1
  Hypermagnesemia, increase to Grade 4, n=77 | 1
  Hypernatremia, any grade increase, n=77 | 9
  Hypernatremia, increase to Grade 3, n=77 | 0
  Hypernatremia, increae to Grade 4, n=77 | 0
  Hypocalcemia, any grade increase, n=71 | 30
  Hypocalcemia, increase to Grade 3, n=71 | 1
  Hypocalcemia, increase to Grade 4, n=71 | 0
  Hypoglycemia, any grade increase, n=77 | 12
  Hypoglycemia, increase to Grade 3, n=77 | 0
  Hypoglycemia, increase to Grade 4, n=77 | 1
  Hypokalemia, any grade increase, n=77 | 15
  Hypokalemia, increase to Grade 3, n=77 | 0
  Hypokalemia, increase to Grade 4, n=77 | 0
  Hypomagnesemia, any grade increase, n=77 | 17
  Hypomagnesemia, increase to Grade 3, n=77 | 0
  Hypomagnesemia, increase Grade 4, n=77 | 0
  Hyponatremia, any grade increase, n=77 | 29
  Hyponatremia, increase to Grade 3, n=77 | 6
  Hyponatremia, increase to Grade 4, n=77 | 0
  Phosphate, any grade increase, n=77 | 32
  Phosphate, increase to Grade 3, n=77 | 3
  Phosphate, increase to Grade 4, n=77 | 0
  TB, any grade increase, n=77 | 40
  TB, increase to Grade 3, n=77 | 4
  TB, increase to Grade 4, n=77 | 0

6. Primary Outcome: Number of Participants With the Indicated Worst-case Grade Increase From Baseline for the Indicated Hematology Parameters at Any Time Post-Baseline
Description: Hematology parameters were summarized according to NIH CTCAE, version 4.0. Grade 1, mild; Grade 2, moderate; Grade 3, severe; Grade 4, life-threatening or disabling; Grade 5, death. Data are presented for only those parameters for which an increase from Baseline occurred. Hematology parameters included: hemoglobin (anemia), lymphocytes (lymphocytopenia), neutrophils (neutropenia), platelets (thrombocytopenia), white blood cells (WBC [leukopenia]), and prothrombin time international normalized ratio (PT [INR]). Participants with missing Baseline grades are assumed to have a Baseline grade of 0.
Time Frame: From Baseline to investigational product discontinuation (up to 6.230 years)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants
  Hemoglobin, any grade increase, n=78 | 29
  Hemoglobin, increase to Grade 3, n=78 | 2
  Hemoglobin, increas to Grade 4, n=78 | 0
  INR (PT), any grade increase, n=67 | 10
  INR (PT), increase to Grade 3, n=67 | 2
  INR (PT), increase to Grade 4, n=67 | 0
  Lymphocytes, any grade increase, n=78 | 34
  Lymphocytes, increase to Grade 3, n=78 | 7
  Lymphocytes, increase to Grade 4, n=78 | 2
  Neutrophils, any grade increase, n=78 | 29
  Neutrophils, increase to Grade 3, n=78 | 1
  Neutrophils, increase to Grade 4, n=78 | 1
  Platelets, any grade increase, n=78 | 31
  Platelets, increase to Grade 3, n=78 | 1
  Platelets, increase to Grade 4, n=78 | 0
  WBC, any grade increase, n=78 | 32
  WBC, increase to Grade 3, n=78 | 2
  WBC, increase to Grade 4, n=78 | 0

7. Primary Outcome: Number of Participants With the Indicated Shift From Baseline in Blood Pressure at Any Time Post-Baseline
Description: Blood pressure measurements included systolic blood pressure (SBP, millimeters of mercury [mmHg]) and diastolic BP (DBP). The number of participants with a post-Baseline shift from Baseline in blood pressure (<90 mmHg, 90 to 139 mmHg, 140 to 169 mmHg, >=170 mmHg) was assessed.
Time Frame: From Baseline to investigational product discontinuation (up to 6.230 years)
Population: ATS Population
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants
  SBP, <90 mmHg | 1
  SBP, 90 to 139 mmHg | 29
  SBP, 140 to 169 mmHg | 44
  SBP, >=170 mmHg | 6
  DBP, <90 mmHg | 1
  DBP, 90 to 139 mmHg | 32
  DBP, 140 to 169 mmHg | 46
  DBP, >=170 mmHg | 1

8. Primary Outcome: Number of Participants With the Indicated Shift in Heart Rate From Baseline at Any Time Post-Baseline
Description: Heart rate is the measure of heart beats per minute (bpm). The number of participants with a post-Baseline shift from Baseline in heart rate of <44 bpm, 44 to 100 bpm, 101 to 120 bpm, and >120 bpm was assessed.
Time Frame: From Baseline to investigational product discontinuation (up to 6.230 years)
Population: ATS Population. Only those participants available at the specified time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 79
participants
  Heart rate <44 bpm | 0
  Heart rate 44 to 100 bpm | 66
  Heart rate 101 to 120 bpm | 12
  Heart rate>120 bpm | 1

9. Primary Outcome: Number of Participants With a Change From Baseline to the Indicated Worst-case Post-Baseline Bazett's Heart Rate-corrected QT Interval (QTc) Value
Description: The QT interval is a measure of the time between the start of the Q wave and the end of the T wave in the heart's electrical cycle. A lengthened QT interval can be a biomarker for ventricular tachyarrhythmias. The QT interval corrected for heart rate using Bazett's formula (QTcB) was calculated; the faster the heart rate, the shorter the QT interval. Electrocardiogram values (Bazett's QTc value) were summarized using the following reference ranges: <450, 450 to 479, 480 to 499, 500 to 549, and >550 milliseconds.
Time Frame: From Baseline to investigational product discontinuation (up to 6.230 years)
Population: ATS Population. Only those participants available at the specified time points were analyzed; 3 participants did not have post-Baseline results.
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 77
participants
  Remained or reduced to <450 | 63
  Remained at Baseline level of 450-479 | 2
  Increased to 450-479 | 8
  Increased to 480-499 | 3
  Increased to >=500 | 1

10. Secondary Outcome: Number of Participants With a Complete Response (CR) or Partial Response (PR)
Description: Overall tumor response is defined as the number of participants achieving either a confirmed complete or partial tumor response per Response Evaluation Criteria in Solid Tumors (RECIST). RECIST guidelines were used to evaluate the measurability of tumor lesions, to determine target and non-target lesions at Baseline, and to evaluate tumor response or disease progression after study start. CR is defined as the disappearance of all target and non-target lesions, and PR is defined as at least a 30% decrease in the sum of the longest diameters (LD) of target lesions, taking as a reference the Baseline sum LD, as assessed by the investigator. Confirmation of a CR/PR required a subsequent assessment of the same response or better at least 28 days after the original response.
Time Frame: From Baseline to Week 24/investigational product discontinuation (up to 3.460 years)
Population: ATS Population
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants
  CR | 0
  PR | 30
  CR+PR | 30

11. Secondary Outcome: Number of Participants With a Response of Confirmed CR+PR+6-month Stable Disease (SD)
Description: The number of participants who achieved either a CR, a PR, or a best response of SD that occurred at least 6 months after screening per RECIST criteria was assessed. CR is defined as the disappearance of all target and non-target lesions; PR is defined as at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the Baseline sum LD; and SD is defined as neither sufficient shrinkage in target lesions to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started and the persistence of one or more non-target lesion(s), as assessed by the investigator. Confirmation of a CR/PR required a subsequent assessment of the same response or better at least 28 days after the original response. A confirmed response of SD required that the SD assessment occurred no earlier than 12 weeks after the screening scans.
Time Frame: From the Baseline to Week 24/investigational product discontinuation (up to 1.65 years)
Population: ATS Population. An analysis was performed on 71 participants.
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 71
participants | 35

12. Secondary Outcome: Number of Participants With the Indicated Best Overall Response
Description: The best overall response is defined as the best response recorded from the start of the treatment until disease progression (PD)/recurrence. Per RECIST: CR, the disappearance of all target and non-target lesions; PR, at least a 30% decrease in the sum of the LD of target lesions, taking as a reference the Baseline sum LD; SD, neither sufficient shrinkage in target lesions to qualify for PR, nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started and the persistence of one or more non-target lesion(s); PD, at least a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum of the LD recorded since the treatment started or the appearance of >=1 new lesion and/or unequivocal progression of existing non-target lesions. Unknown/not evaluable is used for those participants who cannot be classified as achieving CR, PR, SD, or PD.
Time Frame: From the Baseline to Week 24/investigational product discontinuation (up to 3.460 years)
Population: ATS Population
Measure: Number; unit: participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
participants
  Complete Response | 0
  Partial Response | 30
  Stable Disease | 31
  Progressive Disease | 10
  Unknown/Not Evaluable | 9

13. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the interval between the date of the first dose of study medication and the date of disease progression as defined by the investigator or death due to any cause. RECIST was used to evaluate the measurability of tumor lesions, to determine target and non-target lesions at Baseline, and to evaluate tumor response or disease progression after study start. Per RECIST, PD is defined as at least a 20% increase in the sum of the LD of target lesions, taking as a reference the smallest sum of the LD recorded since the treatment started or the appearance of >=1 new lesion and/or unequivocal progression of existing non-target lesions. Participants who did not have disease progression or did not die were censored at the follow-up visit as either follow-up ended or follow-up ongoing. Participants who received non-study anti-cancer therapies before disease progression were treated as censored.
Time Frame: From the first dose of study medication to the earliest date of disease progression (PD) or death due to any cause (up to 3.460 years)
Population: ATS Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
months | 9.2 [7.3 to 12.0]

14. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the interval between the date of the first dose of study medication to the date of death due to any cause. For participants who did not die, time to death was censored at the time of last contact. The last date of contact was defined as the maximum date of any visit date or the survival follow-up date.
Time Frame: as for outcome 13
Population: ATS Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
months | 23.5 [16.3 to 28.0]

15. Secondary Outcome: Percentage of Participants Who Survived Until Month 12
Description: For participants who did not die, time to death was censored at the time of last contact. The last date of contact was defined as the maximum date of any visit date or the survival follow-up date.
Time Frame: From the first dose of study medication to Month 12
Population: ATS Population
Measure: Number; unit: Percentage of participants
Arm/Group | Pazopanib 800 mg
Number analyzed (Participants) | 80
Percentage of participants | 72

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study medication to the end of the treatment period (up to 6.230 years).
Arm/Group | Pazopanib 800 mg
Serious Adverse Events (participants affected / at risk) | 27/80
Other Adverse Events (participants affected / at risk) | 72/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=80)
Pain (General disorders) | 2
Sudden death (General disorders) | 2
Asthenia (General disorders) | 1
Oedema peripheral (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Bone abscess (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cholangitis acute (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Jaundice cholestatic (Hepatobiliary disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Brachial plexopathy (Nervous system disorders) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Cataract (Injury, poisoning and procedural complications) | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 800 mg (N=80)
Diarrhoea (Gastrointestinal disorders) | 35
Nausea (Gastrointestinal disorders) | 20
Abdominal pain (Gastrointestinal disorders) | 15
Vomiting (Gastrointestinal disorders) | 15
Stomatitis (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Hair colour changes (Skin and subcutaneous tissue disorders) | 35
Alopecia (Skin and subcutaneous tissue disorders) | 12
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 7
Hypertension (Vascular disorders) | 35
Fatigue (General disorders) | 15
Asthenia (General disorders) | 9
Chest pain (General disorders) | 7
Mucosal inflammation (General disorders) | 6
Pain (General disorders) | 4
Alanine aminotransferase increased (Investigations) | 12
Aspartate aminotransferase increased (Investigations) | 10
Weight decreased (Investigations) | 10
Blood thyroid stimulating hormone increased (Investigations) | 6
Blood bilirubin increased (Investigations) | 5
Blood lactate dehydrogenase increased (Investigations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 24
Headache (Nervous system disorders) | 13
Dysgeusia (Nervous system disorders) | 10
Dizziness (Nervous system disorders) | 5
Back pain (Musculoskeletal and connective tissue disorders) | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Proteinuria (Renal and urinary disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Hypothyroidism (Endocrine disorders) | 8
Nasopharyngitis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 4
Insomnia (Psychiatric disorders) | 6
Anaemia (Blood and lymphatic system disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.